CLINICAL TRIAL: NCT07094568
Title: Comparative Investigation of Changes in Body Composition and Bone Turnover Markers in People With Obesity After Treatment With Tirzepatide Versus Liraglutide. A Prospective Cohort Study.
Brief Title: Tirzepatide vs Liraglutide in Bone
Acronym: TiLi-BONE
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Laikο General Hospital, Athens (Other); Athens Medical Center (Other); Sotiria General Hospital (Other); 251 Hellenic Air Force & VA General Hospital (Other); Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Maria Yavropoulou, Consultant Endocrinologist in the 1st Department of Propaedeutic and Internal Medicine, Medical School of the National and Kapodistrian University of Athens (NKUA) and Deputy in Charge of (C.E.R.E.D) - Disorders of Calcium and Phosphate Metabolism, National and Kapodistrian University of Athens
Other Study IDs: 7130/23-05-25
Record Dates: First submitted 2025-06-30; First posted 2025-07-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity (Disorder)
Keywords: obesity; bone metabolism; body composition; lean mass; free fat mass; fat mass; tirzepatide; liraglutide; CTX; P1NP
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liraglutide: Patients with obesity receiving liraglutide (up to maximum dose of 3mg daily)
- Tirzepatide: Patients with obesity receiving tirzepatide (up to dose of 10-15mg weekly)

SUMMARY:
This prospective cohort study investigates the effects of tirzepatide versus liraglutide on bone turnover markers and body composition in adults with class 3 obesity, characterised by Body Mass Index (BMI) ≥40 kg/m². Participants will be followed for 6 months with assessments at baseline, 3 and 6. The primary outcome is the change in bone resorption marker C-terminal telopeptide of type I collagen (CTX) at 3 months. Secondary outcomes include changes in body weight, BMI, bone mineral density (BMD), and body composition. The study aims to clarify the differential impact of weight loss achieved through tirzepatide versus liraglutide on bone metabolism and body composition in adults with obesity.

DETAILED DESCRIPTION:
Title of the study Comparative investigation of changes in body composition and bone turnover markers in people with obesity after treatment with tirzepatide versus liraglutide. A prospective cohort study.

Research Hypothesis:

The investigators hypothesize that treatment with tirzepatide versus liraglutide will yield distinct effects on markers of bone turnover and body composition, independent of the magnitude of weight loss due to different molecular mechanisms of action.

Keywords Obesity, Bone Metabolism, Body Composition, Lean mass, Free Fat Mass, Fat Mass, Tirzepatide, Liraglutide, CTX, P1NP, TRAP5b

Introduction Obesity is a growing global health concern, associated with various metabolic disorders, including hypertension, diabetes, metabolic syndrome, non-alcoholic fatty liver disease, sleep apnea and ultimately cardiovascular events. Obesity has also been linked to osteoporosis and high risk of fragility fractures. However, this relationship remains complex, as it involves multiple factors, including mechanical load from body weight, the type and distribution of adipose tissue, imbalances in nutrient intake, and a wide variety of cytokines (adipokines) and hormones secreted by the adipose tissue. On the other hand, rapid and substantial weight loss is associated with a significant reduction in bone mineral density (BMD), osteomalacia and increased risk of fragility fractures. Assessment of bone turnover status can be reliably assessed by circulating levels of bone turnover markers (BTMs) such as the bone resorption markers C-terminal telopeptide of type I (CTX), and tartrate-resistant acid phosphatase (TRAP5b), which evaluates bone resorptive capacity and is not influenced by renal clearance and bone formation markers such as procollagen type 1 N-terminal propeptide (P1NP). Clinical trials have demonstrated that diet-induced weight loss is associated with deterioration of bone metabolism, as indicated by alterations in BTMs and Dual-energy X-ray Absorptiometry (DXA) measurements of BMD. In addition, bariatric management of obesity, particularly malabsorptive surgical modalities, are known to increase the risk of fractures at two years postoperatively. Weight-loss treatments such as liraglutide, the first injectable Glucagon-like peptide-1 (GLP-1) receptor agonist approved for obesity, and tirzepatide, a dual GLP-1/Glucose-dependent insulinotropic polypeptide (GIP) receptor agonist recently approved by the U.S. Food and Drug Administration (FDA) and the European Medicines Agency for treating obesity, has shown efficacy in weight management but their effects on bone metabolism are not fully understood. Liraglutide administration in diabetic mice improves bone health, by altering the levels of BTMs CTX, osteoprotegerin (OPG), osteocalcin (OC), alkaline phosphatase (ALP), and procollagen type 1 N-terminal propeptide (P1NP), reducing the number of osteoclasts, and improving bone architecture. Similarly, in mice models with glucocorticoid-induced osteoporosis (GIOP) under liraglutide treatment, BMD and bone microarchitecture is improved, with reductions in BTMs such as Tartrate-resistant acid phosphatase type 5b (TRACP-5b) and CTX, and increases in ALP and OPG. A randomized, double-blinded, placebo-controlled clinical trial of 56 individuals with diabetes (mean age: 63 years) showed that liraglutide at a dose of 1.8 mg did not affect bone metabolism despite a reduction in body weight. Another randomized controlled study of 37 women with obesity (mean age 46 years, BMI 34kg/m2) who lost 12% of body weight after a 12-week low-calorie diet and were subsequently randomized to placebo or liraglutide at a dose of 1.2 mg, found that liraglutide increased P1NP levels by 16%, highlighting its positive effects on bone metabolism following weight loss. Nevertheless, clinical data on the effects of liraglutide on bone metabolism are limited. Regarding tirzepatide, the pronounced weight loss from its administration seems to have a neutral effect on bone mass and microarchitecture in diabetic mice, with no significant changes in BTMs. However, no clinical data are currently available regarding tirzepatide effect on bone metabolism. The concern, however, is that the combination of GLP-1 and GIP, which leads to greater weight loss, may have a different impact on bone metabolism than GLP-1 agonists alone.

Necessity/ Originality The available human studies in populations with diabetes and obesity are limited, with most reaching a maximum dose of Liraglutide in 1.8 mg daily and not resulting in significant weight loss associations with bone metabolism. There are no human studies with tirzepatide concerning its impact on bone metabolism.

The necessity and originality of the study lies in the fact that no previous research has investigated the effects of tirzepatide (at maximum doses of 10 -15 mg weekly) and liraglutide (at dose of 3 mg daily) on both body composition parameters and bone metabolism in individuals with obesity.

The aim of the present study is to investigate the potential differential effects of tirzepatide versus liraglutide on bone turnover status and body composition parameters in patients living with obesity and explore the association with differences in the magnitude of weight loss and the different mechanisms of action (GlP-1 agonism versus GIP/GLP-1 synergy).

Primary - Objectives:

1. To evaluate the impact of tirzepatide on bone turnover status and bone mineral density in patients with obesity.
2. To assess the effects of liraglutide on bone turnover status and bone mineral density in patients with obesity.
3. To compare the alterations in bone metabolism across the 2 intervention groups, after adjustments for the differences in weight loss.

Secondary - Objectives:

1. To evaluate the impact of tirzepatide on body composition parameters in patients with obesity.
2. To assess the effects of liraglutide on body composition parameters in patients with obesity.
3. To compare the alterations in body composition parameters across the 2 intervention groups, after adjustments for the differences in weight loss.

Significance of the Study/ Clinical relevance This research will provide valuable data regarding the effects of weight-loss medications on bone health and body composition in individuals living with obesity. The findings may influence clinical practice guidelines and therapeutic approaches in managing obesity and its associated complications.

Methodology

1. Study Design:

   Open-label observational cohort study
2. Inclusion Criteria-Participants:

   Adults aged over 30 years with BMI ≥40 kg/m²
3. Exclusion criteria:

   * Type 2 Diabetes Mellitus (T2DM) and type 1 Diabetes Mellitus (T1DM)
   * Chronic kidney disease
   * Liver failure
   * Heart failure
   * Malignancy coexistence
   * Previous bariatric or gastrointestinal surgery involving intestinal bypass
   * Uncontrolled hypo/hyperthyroidism
   * Uncontrolled hypo/hyperparathyroidism
   * Pregnancy and lactation
   * Recent fracture (within 2 years)
   * Rare Metabolic Bone Diseases (e.g., Paget's disease of bone, fibrous dysplasia, osteopetrosis)
   * Inflammatory arthritis
   * Medications which can affect bone markers: bone-anabolic agents, antiresorptive agents, antiandrogenic agents, vitamin K antagonists, antipsychotic agents, contraceptives, glucocorticoids (oral), methotrexate, thiazides, aromatase inhibitors etc)
   * Hemolytic anemia

   Patients who will be deemed eligible for the study and sign the informed consent form will undergo the following research protocol.
4. The step-by-step process of the study Visit 1 Medical history documentation and measurement of anthropometric parameters (Height, Weight, BMI, Waist-to-Hip Ratio, waist to height ratio).

   Assessment of SARC-F questionnaire , Short-Form 36 (SF-36) Health Survey and Perceived Stress Scale - 14 item (PSS-14) (validated for the Greek population).

   Bioelectrical impedance analysis (BIA) Resting Metabolic Rate (RMR). Grip strength, Chair stand test and Gait speed. DXA at three skeletal sites (lumbar spine and both hips), calculation of Trabecular Bone Score (TBS) and Whole-Body Scan.

   Blood sampling*. Hypocaloric diet designed by the same dietary team, providing an energy intake 20-30% below the Total Energy Expenditure, as estimated from the Resting Metabolic Rate and exercise recommendations.

   Patients then will be prescribed liraglutide or tirzepatide based on their discretion and their treating physician's choice.

   Weekly estimation of each participant from Group A - liraglutide Group to assess the potential for a dosage increase starting from an initial dose of 0.6 mg daily, with incremental increases of 0.6 mg, up to the maximum tolerated dose, with a maximum target dose of 3 mg per day.

   Monthly estimation of each patient from Group B - tirzepatide Group to assess the potential for a dosage increase, starting from an initial dose of 2.5 mg weekly, up to the maximum tolerated dose, with a maximum target dose of 10-15 mg per week.

   Visit 2-Follow up in 3rd month Medical history documentation and measurement of anthropometric parameters (Height, Weight, BMI, Waist-to-Hip Ratio, waist to height ratio).

   BIA. Grip strength, Chair stand test and Gait speed. Blood sampling*. Patients continue to receive liraglutide or tirzepatide. Monitoring the adherence to the diet and exercise program based on the patient's reports.

   Visit 3-Follow up in 6th month Medical history documentation and measurement of anthropometric parameters (Height, Weight, BMI, Waist-to-Hip Ratio, waist to height ratio).

   Assessment of SARC-F questionnaire, SF-36 Health Survey and PSS-14 (35) (validated for the Greek population).

   BIA. RMR. Grip strength, Chair stand test and Gait speed. DXA at three skeletal sites (lumbar spine and both hips), calculation of TBS and Whole-Body Scan.

   Blood sampling*. Patients continue to receive liraglutide or tirzepatide. Monitoring the adherence to the diet and exercise program based on the patient's reports.

   * Blood sampling for the determination of CTX, P1NP, TRAPC5b, OC, calcium, phosphate, albumin, ALP, parathyroid hormone (PTH), 25-hydroxyvitamin D [25(OH)D], insulin-like growth factor 1 (IGF1), adiponectin, leptin, and insulin will be conducted during the morning hours between 8 and 10 a.m., following an 8-hour fasting period and avoidance of strenuous exercise the previous day. For premenopausal women, blood sampling will be conducted during the follicular phase of the menstrual cycle, based on the patient's menstrual history.
5. Study Endpoints:

   * The primary endpoint is to investigate comparative changes in the bone resorption marker CTX at 3 months with liraglutide vs tirzepatide.
   * Secondary endpoints include:

     1. changes in body weight and BMI at 6 months
     2. BMD and body composition parameters measured by DXA scan at baseline and after 6 months of intervention.
6. Data Analysis:

   * Statistical analysis will be performed using ANOVA for comparison between groups. Correlation with changes in weight and bone metabolism indices will also be assessed using regression analysis.
7. Sample size calculation The sample size calculation for this study was based on the least significant change (LSC) of the C-terminal telopeptide of type I collagen (CTX) marker in serum at three months. Using this threshold, the investigators determined that a total of 32 patients per arm would be required to achieve adequate statistical power (80% statistical power (false negative), 5% error (false positive). With anticipated drop-out rate of 10%, about 36 participants/ per group should be randomized, ensuring sufficient power to detect meaningful changes in CTX levels while accounting for potential variability in the biomarker response.
8. Recruitment centers Laikο General Hospital, Athens Athens Medical Center Sotiria General Hospital 251 Hellenic Air Force & VA General Hospital Evangelismos Hospital
9. Protocol for Sample Collection and Processing Fasting Status: Blood samples are collected after an overnight fast. Vigorous exercise is avoided on the day prior to sample collection.

   Timing of Collection: Samples are collected between 7:30 a.m. and 10:00 a.m. Sample Type: Serum and EDTA plasma are used. Sample Processing: Samples are centrifuged immediately and serum and plasma separated and stored into aliquots. Hemolysis is avoided during handling.

   Storage Conditions: Samples are stored at ≤-20 °C until analysis. For long-term storage exceeding three months for CTX-I and six months for PINP, samples are maintained at ≤-70 °C.

   Thawing and Preparation: Thawed samples are mixed thoroughly by inversion before analysis. Centrifugation is performed to remove particulates when necessary.

   Consistency in Monitoring: The same sample type and identical handling conditions are maintained for patient monitoring.

   Batch Analysis of Serial Samples: Serial samples are frozen and analyzed collectively within the same batch.
10. Ethics The study will be reviewed and approved by the Ethics Committee of LAIKO General Hospital of Athens and the Ethics Committee of the Medical School of National and Kapodistrian University of Athens, before initiation. It will be conducted in compliance with the ethical principles outlined in the Declaration of Helsinki, ensuring the protection of participants' rights, safety, and well-being. All participants will provide informed consent before enrollment, and the study will adhere to all relevant regulatory and institutional guidelines for clinical research.
11. Processing capabilities:

1. Timeline: Recruitment: 6 months; may be extended up to 12 months Data Analysis: 3 months Authorship: at least 2 years

2. Budget: A detailed budget will be prepared, covering personnel costs, laboratory tests, participant incentives, and data analysis.

Conclusion:

This research aims to fill the gap in knowledge regarding how different interventions for obesity affect bone metabolism, which is crucial for developing comprehensive treatment protocols for people living with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 30 and 65 years
* BMI ≥40 kg/m²

Exclusion Criteria:

* Type 2 Diabetes Mellitus (T2DM) and type 1 Diabetes Mellitus (T1DM)
* Chronic kidney disease
* Liver failure
* Heart failure
* Malignancy coexistence
* Previous bariatric or gastrointestinal surgery involving intestinal bypass
* Uncontrolled hypo/hyperthyroidism
* Uncontrolled hypo/hyperparathyroidism
* Pregnancy and lactation
* Recent fracture (within 2 years)
* Rare Metabolic Bone Diseases (e.g., Paget's disease of bone, fibrous dysplasia, osteopetrosis)
* Inflammatory arthritis
* Medications which can affect bone markers: bone-anabolic agents, antiresorptive agents, antiandrogenic agents, vitamin K antagonists, antipsychotic agents, contraceptives, glucocorticoids (oral), methotrexate, thiazides, aromatase inhibitors etc)
* Hemolytic anemia

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves patients with a body mass index (BMI) greater than 40 who either present for weight loss management at endocrinology or obesity clinics, or who are referred to sleep disorder centers due to obstructive sleep apnea syndrome requiring CPAP therapy, where weight loss intervention is consequently recommended.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum CTX concentration | Baseline and 3 months after intervention initiation
  Evaluation of changes in the bone resorption marker CTX at 3 months after intervention initiation in participants treated with tirzepatide versus liraglutide

SECONDARY OUTCOMES:
Change in body weight | Baseline and 6 months after intervention initiation
  Evaluation of changes in body weight at 6 months after intervention initiation in participants treated with tirzepatide versus liraglutide
Change in Body Mass Index (BMI) | Baseline and 6 months after intervention initiation
  Evaluation of changes in BMI at 6 months after intervention initiation in participants treated with tirzepatide versus liraglutide
Change in Bone Mineral Density (BMD) | Baseline and 6 months after intervention initiation
  Evaluation of changes in BMD measured by DXA scan at 6 months after intervention initiation in participants treated with tirzepatide versus liraglutide
Change in Body Composition Parameters | Baseline and 6 months after intervention initiation
  Evaluation of changes in android fat mass, gynoid fat mass, android-to-gynoid fat ratio, trunk-to-legs fat percentage ratio, trunk-to-limb fat mass ratio, appendicular lean mass index and total fat mass measured by DXA whole-body scan at baseline and 6 months after intervention initiation in participants treated with tirzepatide versus liraglutide

CONTACTS AND LOCATIONS:
Locations (1):
- Laiko General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Due to participant privacy concerns and institutional policies, individual participant data will not be shared outside the research team

REFERENCES:
- [Result] Greenblatt MB, Tsai JN, Wein MN. Bone Turnover Markers in the Diagnosis and Monitoring of Metabolic Bone Disease. Clin Chem. 2017 Feb;63(2):464-474. doi: 10.1373/clinchem.2016.259085. Epub 2016 Dec 9. PMID 27940448
- [Result] Katsarou A, Panagiotakos D, Zafeiropoulou A, Vryonis M, Skoularigis I, Tryposkiadis F, Papageorgiou C. Validation of a Greek version of PSS-14; a global measure of perceived stress. Cent Eur J Public Health. 2012 Jun;20(2):104-9. doi: 10.21101/cejph.a3698. PMID 22966732
- [Result] Pappa E, Kontodimopoulos N, Niakas D. Validating and norming of the Greek SF-36 Health Survey. Qual Life Res. 2005 Jun;14(5):1433-8. doi: 10.1007/s11136-004-6014-y. PMID 16047519
- [Result] Tsekoura M, Billis E, Tsepis E, Lampropoulou S, Beaudart C, Bruyere O, Yilmaz O, Bahat G, Gliatis J. Cross-cultural adaptation and validation of the Greek Version of the SARC-F for evaluating sarcopenia in Greek older adults. J Musculoskelet Neuronal Interact. 2020 Dec 1;20(4):505-512. PMID 33265078
- [Result] Denarie D, Constant E, Thomas T, Marotte H. Could biomarkers of bone, cartilage or synovium turnover be used for relapse prediction in rheumatoid arthritis patients? Mediators Inflamm. 2014;2014:537324. doi: 10.1155/2014/537324. Epub 2014 Mar 12. PMID 24744505
- [Result] Farup PG. Changes in bone turnover markers 6-12 months after bariatric surgery. Sci Rep. 2024 Jun 27;14(1):14844. doi: 10.1038/s41598-024-65952-y. PMID 38937532
- [Result] Wu C, Kato TS, Pronschinske K, Qiu S, Naka Y, Takayama H, Schulze-Spate U, Cremers S, Shane E, Mancini D, Schulze PC. Dynamics of bone turnover markers in patients with heart failure and following haemodynamic improvement through ventricular assist device implantation. Eur J Heart Fail. 2012 Dec;14(12):1356-65. doi: 10.1093/eurjhf/hfs138. Epub 2012 Sep 18. PMID 22989867
- [Result] Woodcock A. Effects of inhaled corticosteroids on bone density and metabolism. J Allergy Clin Immunol. 1998 Apr;101(4 Pt 2):S456-9. doi: 10.1016/s0091-6749(98)70159-9. PMID 9563372
- [Result] Weerasinghe DK, Hodge JM, Pasco JA, Samarasinghe RM, Azimi Manavi B, Williams LJ. Antipsychotic-induced bone loss: the role of dopamine, serotonin and adrenergic receptor signalling. Front Cell Dev Biol. 2023 May 25;11:1184550. doi: 10.3389/fcell.2023.1184550. eCollection 2023. PMID 37305679
- [Result] Loncar G, Cvetinovic N, Lainscak M, Isakovic A, von Haehling S. Bone in heart failure. J Cachexia Sarcopenia Muscle. 2020 Apr;11(2):381-393. doi: 10.1002/jcsm.12516. Epub 2020 Feb 22. PMID 32087616
- [Result] Vasikaran S, Eastell R, Bruyere O, Foldes AJ, Garnero P, Griesmacher A, McClung M, Morris HA, Silverman S, Trenti T, Wahl DA, Cooper C, Kanis JA; IOF-IFCC Bone Marker Standards Working Group. Markers of bone turnover for the prediction of fracture risk and monitoring of osteoporosis treatment: a need for international reference standards. Osteoporos Int. 2011 Feb;22(2):391-420. doi: 10.1007/s00198-010-1501-1. Epub 2010 Dec 24. PMID 21184054
- [Result] Schini M, Vilaca T, Gossiel F, Salam S, Eastell R. Bone Turnover Markers: Basic Biology to Clinical Applications. Endocr Rev. 2023 May 8;44(3):417-473. doi: 10.1210/endrev/bnac031. PMID 36510335
- [Result] Filella X, Guanabens N. Clinical use of bone markers: a challenge to variability. Adv Lab Med. 2023 Aug 28;5(1):7-14. doi: 10.1515/almed-2023-0092. eCollection 2024 Mar. PMID 38634081
- [Result] Lv F, Cai X, Lin C, Yang W, Ji L. Effects of Semaglutide and Tirzepatide on Bone Metabolism in Type 2 Diabetic Mice. Pharmaceuticals (Basel). 2024 Dec 9;17(12):1655. doi: 10.3390/ph17121655. PMID 39770498
- [Result] Iepsen EW, Lundgren JR, Hartmann B, Pedersen O, Hansen T, Jorgensen NR, Jensen JE, Holst JJ, Madsbad S, Torekov SS. GLP-1 Receptor Agonist Treatment Increases Bone Formation and Prevents Bone Loss in Weight-Reduced Obese Women. J Clin Endocrinol Metab. 2015 Aug;100(8):2909-17. doi: 10.1210/jc.2015-1176. Epub 2015 Jun 4. PMID 26043228
- [Result] Hygum K, Harslof T, Jorgensen NR, Rungby J, Pedersen SB, Langdahl BL. Bone resorption is unchanged by liraglutide in type 2 diabetes patients: A randomised controlled trial. Bone. 2020 Mar;132:115197. doi: 10.1016/j.bone.2019.115197. Epub 2019 Dec 20. PMID 31870634
- [Result] Yang L, Yang J, Pan T, Zhong X. Liraglutide increases bone formation and inhibits bone resorption in rats with glucocorticoid-induced osteoporosis. J Endocrinol Invest. 2019 Sep;42(9):1125-1131. doi: 10.1007/s40618-019-01034-5. Epub 2019 Apr 6. PMID 30955181
- [Result] Cheng Y, Liu P, Xiang Q, Liang J, Chen H, Zhang H, Yang L. Glucagon-like peptide-1 attenuates diabetes-associated osteoporosis in ZDF rat, possibly through the RAGE pathway. BMC Musculoskelet Disord. 2022 May 17;23(1):465. doi: 10.1186/s12891-022-05396-5. PMID 35581617
- [Result] Wen B, Zhao L, Zhao H, Wang X. Liraglutide exerts a bone-protective effect in ovariectomized rats with streptozotocin-induced diabetes by inhibiting osteoclastogenesis. Exp Ther Med. 2018 Jun;15(6):5077-5083. doi: 10.3892/etm.2018.6043. Epub 2018 Apr 10. PMID 29805533
- [Result] Fathy MA, Anbaig A, Aljafil R, El-Sayed SF, Abdelnour HM, Ahmed MM, Abdelghany EMA, Alnasser SM, Hassan SMA, Shalaby AM. Effect of Liraglutide on Osteoporosis in a Rat Model of Type 2 Diabetes Mellitus: A Histological, Immunohistochemical, and Biochemical Study. Microsc Microanal. 2023 Dec 21;29(6):2053-2067. doi: 10.1093/micmic/ozad102. PMID 37832035
- [Result] Stefanakis K, Kokkorakis M, Mantzoros CS. The impact of weight loss on fat-free mass, muscle, bone and hematopoiesis health: Implications for emerging pharmacotherapies aiming at fat reduction and lean mass preservation. Metabolism. 2024 Dec;161:156057. doi: 10.1016/j.metabol.2024.156057. Epub 2024 Oct 30. PMID 39481534
- [Result] Batsis JA. Obesity in the Older Adult: Special Issue. J Nutr Gerontol Geriatr. 2019 Jan-Mar;38(1):1-5. doi: 10.1080/21551197.2018.1564197. Epub 2019 Feb 26. No abstract available. PMID 30806583
- [Result] Saad RK, Ghezzawi M, Habli D, Alami RS, Chakhtoura M. Fracture risk following bariatric surgery: a systematic review and meta-analysis. Osteoporos Int. 2022 Mar;33(3):511-526. doi: 10.1007/s00198-021-06206-9. Epub 2022 Jan 5. PMID 34988627
- [Result] Wright CS, Li J, Campbell WW. Effects of Dietary Protein Quantity on Bone Quantity following Weight Loss: A Systematic Review and Meta-analysis. Adv Nutr. 2019 Nov 1;10(6):1089-1107. doi: 10.1093/advances/nmz058. PMID 31301138
- [Result] Zibellini J, Seimon RV, Lee CM, Gibson AA, Hsu MS, Shapses SA, Nguyen TV, Sainsbury A. Does Diet-Induced Weight Loss Lead to Bone Loss in Overweight or Obese Adults? A Systematic Review and Meta-Analysis of Clinical Trials. J Bone Miner Res. 2015 Dec;30(12):2168-78. doi: 10.1002/jbmr.2564. Epub 2015 Jun 16. PMID 26012544
- [Result] Szulc P, Naylor K, Hoyle NR, Eastell R, Leary ET; National Bone Health Alliance Bone Turnover Marker Project. Use of CTX-I and PINP as bone turnover markers: National Bone Health Alliance recommendations to standardize sample handling and patient preparation to reduce pre-analytical variability. Osteoporos Int. 2017 Sep;28(9):2541-2556. doi: 10.1007/s00198-017-4082-4. Epub 2017 Jun 19. PMID 28631236
- [Result] Patel N, Ganti L. The Treatment and Monitoring of Osteoporosis using Bone Turnover Markers. Orthop Rev (Pavia). 2025 Jan 6;17:127772. doi: 10.52965/001c.127772. eCollection 2025. PMID 39790440
- [Result] Hunter GR, Plaisance EP, Fisher G. Weight loss and bone mineral density. Curr Opin Endocrinol Diabetes Obes. 2014 Oct;21(5):358-62. doi: 10.1097/MED.0000000000000087. PMID 25105997
- [Result] Rinonapoli G, Pace V, Ruggiero C, Ceccarini P, Bisaccia M, Meccariello L, Caraffa A. Obesity and Bone: A Complex Relationship. Int J Mol Sci. 2021 Dec 20;22(24):13662. doi: 10.3390/ijms222413662. PMID 34948466
- [Result] Li H, Qiu J, Gao Z, Li C, Chu J. Association between waist-to-height ratio and osteoporosis in the National Health and Nutrition Examination Survey: a cross-sectional study. Front Med (Lausanne). 2024 Dec 18;11:1486611. doi: 10.3389/fmed.2024.1486611. eCollection 2024. PMID 39744530
- [Result] Liu Y, Liu Y, Huang Y, Le S, Jiang H, Ruan B, Ao X, Shi X, Fu X, Wang S. The effect of overweight or obesity on osteoporosis: A systematic review and meta-analysis. Clin Nutr. 2023 Dec;42(12):2457-2467. doi: 10.1016/j.clnu.2023.10.013. Epub 2023 Oct 18. PMID 37925778
- [Result] Hou J, He C, He W, Yang M, Luo X, Li C. Obesity and Bone Health: A Complex Link. Front Cell Dev Biol. 2020 Dec 21;8:600181. doi: 10.3389/fcell.2020.600181. eCollection 2020. PMID 33409277
- [Result] Gkastaris K, Goulis DG, Potoupnis M, Anastasilakis AD, Kapetanos G. Obesity, osteoporosis and bone metabolism. J Musculoskelet Neuronal Interact. 2020 Sep 1;20(3):372-381. PMID 32877973
- [Result] Cauley JA. Public health impact of osteoporosis. J Gerontol A Biol Sci Med Sci. 2013 Oct;68(10):1243-51. doi: 10.1093/gerona/glt093. Epub 2013 Jul 31. PMID 23902935
- [Result] Rhee EJ. The Influence of Obesity and Metabolic Health on Vascular Health. Endocrinol Metab (Seoul). 2022 Feb;37(1):1-8. doi: 10.3803/EnM.2022.101. Epub 2022 Feb 28. PMID 35255597
- [Result] Engin A. The Definition and Prevalence of Obesity and Metabolic Syndrome. Adv Exp Med Biol. 2017;960:1-17. doi: 10.1007/978-3-319-48382-5_1. PMID 28585193